CLINICAL TRIAL: NCT01108484
Title: Evaluation of the Effects of Exercise, Diet and Control of Psychological Stress in Cancer Survivors
Brief Title: Program of Exercise, Diet and Control of Psychological Stress in Cancer Survivors
Acronym: EDICOS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Grupo de Investigación en Actividad Física y Salud (Other)
Responsible Party: Principal Investigator, Fernando Herrero, MD PhD, Grupo de Investigación en Actividad Física y Salud
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: GIAFYS-2010-01
Record Dates: First submitted 2010-04-20; First posted 2010-04-22 (Estimated); Last update posted 2020-11-30 (Actual); Status verified 2020-11

CONDITIONS: Cancer Survivors
Keywords: Cancer survivors, exercise, diet, emotional support
MeSH Terms: conditions — Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Supervised exercise (Experimental): Cardiorespiratory and resistance training
  Interventions: Behavioral: Exercise
- Exercise + diet counseling (Experimental): Cardiorespiratory and resistance training + Diet counseling to improve food intake(more fruit and vegetable and less fat food)
  Interventions: Behavioral: Exercise + Diet counseling
- Exercise + diet counseling + psycho support (Experimental): Cardiorespiratory and resistance training + Diet counseling to improve food intake(more fruit and vegetable and less fat food) + Weekly sessions to modify the behaviour
  Interventions: Behavioral: Exercise + Diet counseling + psycho-emotional support
- Control (No Intervention): They will keep their usual way of life

INTERVENTIONS:
Behavioral: Exercise — Supervised exercise: Three 90-minutes sessions per week.
  Arms: Supervised exercise
Behavioral: Exercise + Diet counseling — Supervised exercise: Three 90-minutes sessions per week. Diet counseling: Counseling to balance the intake.
  Arms: Exercise + diet counseling
Behavioral: Exercise + Diet counseling + psycho-emotional support — Supervised exercise: Three 90-minutes sessions per week. Diet counseling: Counseling to balance the intake. Psycho-emotional support: Weekly sessions to modify the behaviour.
  Arms: Exercise + diet counseling + psycho support

SUMMARY:
A program of exercise, diet and psycho-emotional support could improve some outcomes in cancer survivors.

DETAILED DESCRIPTION:
Cancer survivors will be randomised to one of the following groups: a) Supervised physical activity, b) Supervised physical activity + Diet counseling, c) Supervised physical activity + Diet counseling + psycho-emotional support

ELIGIBILITY:
Inclusion Criteria:

* cancer survivors attending their follow-up visits

Exclusion Criteria:

* Cardiac disease NYHA II
* non-controlled hypertension
* non-controlled metabolic disease
* chronic infectious disease
* non-controlled pain
* risk of bone fracture
* severe anemia, leucopenia or thrombopenia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2010-03; Primary Completion 2015-07 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
VO2 max | basal, 6, 12 and 24 months
  the highest rate of oxygen consumption attainable during maximal exercise

SECONDARY OUTCOMES:
Physical Activity Quality of life Food intake Anxiety and Psychological Distress | basal, 6, 12 and 24 months
  Measured through accelerometer, PAR, CFCA, EORTC QLQ C-30 and SF-36

CONTACTS AND LOCATIONS:
Overall Officials: Fernando Herrero-Roman, MD PhD, Study Chair — Grupo de Investigación en Actividad Física y Salud
Locations (2):
- Spain (2):
  - GIAFYS headquarters, Miranda de Ebro, Burgos
  - GIAFYS, Miranda de Ebro, Burgos